CLINICAL TRIAL: NCT05340946
Title: Comparison of the Effect of Two Anaesthesia Methods in Preventing Perioperative Myocardial Infarction in Patients With Cardiac Risk Undergoing Total Knee Arthroplasty
Brief Title: Comparison of the Effect of Two Anaesthesia Methods in Preventing Perioperative Myocardial Infarcation in Patients With Cardiac Risk Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0305415
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Ischaemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Anesthesia, General; Analgesia, Patient-Controlled; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: The aim of this study is to compare the effect of two anaesthesia methods in preventing perioperative myocardial infarction in patients with cardiac risk undergoing total knee arthroplasty. The primary outcome included perioperative levels of brain natriuretic peptide & cardiac troponins. Secondary outcomes included postoperative operative pain assessment using visual analogue scale, total amount of analgesic consumption, patient satisfaction & cardiovascular complications (myocardial infarction, arrhythmias , heart failure, hypotension, hypertension & the need for inotropic agents ).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (G) (Experimental): received general anaesthesia followed by IV patient-controlled analgesia (IV PCA).
  Interventions: Procedure: general anaesthesia
- Group (F) (Experimental): received spinal anaesthesia followed by continuous ultrasound guided femoral never block once the anaesthesia-induced motor block resolved.
  Interventions: Procedure: spinal anaesthesia

INTERVENTIONS:
Procedure: general anaesthesia — intraoperative general anaesthesia followed by postoperative IV patient analgesia
  Other Names: intravenous patient controlled analgesia
  Arms: Group (G)
Procedure: spinal anaesthesia — patient received spinal followed by continuous ultrasound guided femoral never block.
  Other Names: ultrasound guided femoral never block
  Arms: Group (F)

SUMMARY:
Comparison of the effect of two anaesthesia methods in preventing perioperative myocardial infarction in patients with cardiac risk undergoing total knee arthroplasty

DETAILED DESCRIPTION:
we enrolled 50 patients of both sex of American society of Anesthesiologists (ASA) physical status II where the presence and/or risk for coronary artery disease (CAD) as well as planned lower extremity surgery was considered. Presence of CAD was ascertained by history of myocardial infarction and diagnosis of typical angina or atypical angina with a positive stress test & ECG finding. Risk for CAD included age (> 65 years old), hypertension, smoking habit, blood cholesterol (>240 mg/dL), and diabetes. who met the selection criteria were randomly allocated to 1 of the 2 groups (25 patients) each:

* Group (G): received general anaesthesia followed by IV patient-controlled analgesia (IV PCA).
* Group (F): received spinal anaesthesia followed by continuous ultrasound guided femoral never block once the anaesthesia-induced motor block resolved. We aimed to compare the effect of the two anaesthesia methods in preventing perioperative myocardial infarction in patients with cardiac risk undergoing total knee arthroplasty. The primary outcome included perioperative levels of brain natriuretic peptide & cardiac troponins. Secondary outcomes included postoperative operative pain assessment using visual analogue scale, total amount of analgesic consumption, patient satisfaction & cardiovascular complications (myocardial infarction, arrhythmias , heart failure, hypotension, hypertension & the need for inotropic agents).

ELIGIBILITY:
Inclusion Criteria:

* presence and/or risk for coronary artery disease (CAD) as well as planned lower extremity surgery was considered. Presence of CAD was ascertained by history of myocardial infarction and diagnosis of typical angina or atypical angina with a positive stress test & ECG finding. Risk for CAD included age (> 65 years old), hypertension, smoking habit, blood cholesterol (>240 mg/dL), and diabetes.

Exclusion Criteria:

* 1) severe impairment of left ventricular function (ejection fraction < 40 %). 2) renal failure requiring hemodialysis. 3) known allergies to the drugs used in the present study. 4) contraindications to regional blocks (localized infection, and use of an antiplatelet drug within 3 days before the surgery). 5) unusual blood coagulation tests.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
brain natriuretic peptide | immediately preoperatively
  marker for myocardial infarction
brain natriuretic peptide | after 48 hours post-operatively
  marker for myocardial infarction

SECONDARY OUTCOMES:
visual analogue scale | after 6 hour postoperatively
  a score to evaluate postoperative pain intensity
amount of analgesic consumption | after 48 hour postoperatively
  the total amount of analgesic consumed by each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No